CLINICAL TRIAL: NCT05033587
Title: AK105 With Anlotinib and Radiotherapy Adjuvant Therapy in MGMT Unmethylated Newly Diagnosed Glioblastoma: a Prospective, Open-label Single-arm, Exploratory Trial.
Brief Title: Study of AK105 With Anlotinib and Radiotherapy Adjuvant Therapy in MGMT Unmethylated Newly Diagnosed Glioblastoma.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yang Yang, Professor of medicine, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-252-02
Record Dates: First submitted 2021-08-27; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: MGMT-Unmethylated Glioblastoma
MeSH Terms: interventions — anlotinib; penpulimab; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK105 injection with anlotinib and radiotherapy (Experimental): AK105 200mg intravenously (IV) on day 1 of each 21-day cycle until disease progression or treatment intolerance, the dose can not be adjusted.
  Anlotinib 12mg capsules given orally on once daily in 21-day cycle until disease progression or treatment intolerance(14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21), the dose can be adjusted to 10mg or 8mg according to the specific conditions of the patient.
  The conventional radiotherapy regimen delivered 2.0Gy once a day, five days a week to a total dose of 60Gy.
  Interventions: Drug: Anlotinib; Drug: AK105; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Anlotinib — Anlotinib a multi-target receptor tyrosine kinase inhibitor.
  Other Names: Anlotinib Hydrochloride Capsules
Drug: AK105 — AK105 is a humanized monoclonal antibody that specifically binds to PD-1.
  Other Names: Penpulimab Injection
Radiation: Radiotherapy — The radiotherapy regimen delivered 2.0Gy once a day, five days a week to a total dose of 60Gy.

SUMMARY:
This is a prospective, open-label single-arm, exploratory, two-stage design trial, aiming to investigate safety and efficacy of AK105 with anlotinib and radiotherapy adjuvant therapy in MGMT unmethylated newly diagnosed glioblastoma.

DETAILED DESCRIPTION:
Glioblastoma is the most common and aggressive primary brain tumor in adults. Treatment usually involves surgery, after which chemotherapy and radiation therapy are used. The Central Brain Tumor Registry of the United States (CBTRUS) Statistical Report primary brain and other central nervous system tumors diagnosed in the United States in 2012-2016, glioblastoma accounted for 48.3% of primary malignant brain tumors.

The Stupp protocol has become standard of care for the treatment of newly diagnosed GBM, however, some MGMT unmethylated glioblastomas are still resistant to temozolomide.

Immunotherapy is being studied as treatment for the cancer, AK105 is a humanized monoclonal antibody that specially binds to PD-1. Anlotinib hydrochloride is a multi-target receptor tyrosine kinase inhibitor. Based on the mechanism study, tumor vascular abnormalities promote tissue hypoxia and increase lactic acid, thereby activating immunosuppression and inhibiting T cell function. Anti-angiogenic drugs enhance the infiltration of effector immune cells by inducing normalization of blood vessels and reducing immunosuppression.

ELIGIBILITY:
Inclusion Criteria:

* The patient voluntarily joined the study and signed a written informed consent;
* Pathologically confirmed treatment-naïve glioblastoma with PCR tested MGMT unmethylated;
* The interval between the last biopsy or surgery is 4-6 weeks, and the surgical incision is healed well;
* According to Rano criteria, there are evaluable measurable disease;
* 18-70 years of age;
* Karnofsky performance status (KPS) ≥ 60; and estimated survival of at least 3 months;
* The main organ function to meet the following criteria:

  1) routine blood test: HB≥90g/L(no blood transfusion in 14 days); ANC≥1.5×109/L; White blood cell counts≥3.5×109/L; PLT≥90×109/L; 2) blood biochemical test: ALT and AST ≤2.5×ULN(times the upper limit of normal) and if liver/bone metastases≤5×ULN; TBIL ≤1.5 ULN; Serum Cr≤1.5×ULN and CrCL≥60 ml/min; 3) APTT, INR and PT≤1.5×ULN;
* The woman patients of childbearing age who must agree to take contraceptive methods during the research and within another 6 months after it; who are not in the lactation period and examined as negative in blood serum test or urine pregnancy test within 7 days before the research.

Exclusion Criteria:

* Prior therapy with anti-angiogenic drugs, such as anlotinib, apatinib, lenvatinib, sorafenib, sunitinib, surufatinib, regorafenib or fruquintinib ect, or with anti-PD-1(L1) or anti-CTLA-4 agents;
* Patients who get other monoclonal antibodies have severe hypersensitivity;
* Present or along with other malignancies within 5 years. Exceptions include cured basal cell carcinoma of the skin or in situ prostate cancer or in situ cervical cancer;
* Patients have any active autoimmune disease that required systemic treatment, including but not limited to autoimmune hepatitis, enteritis, vasculitis, nephritis; asthma that require bronchodilators for medical intervention. Exceptions include patients with vitiligo, psoriasis, alopecia or well-controlled type 1 diabetes but not required systemic treatment, or hypothyroidism with normal thyroid function after alternative treatment;
* In the past, there is a treatment toxicity of CTCAE5.0 ≥2 grade that has not been completely relieved (the adverse reaction grades in this article, unless otherwise specified, are defaulted to the CTCAE 5.0 standard);
* Immunodeficiency diagnosis or receiving chronic systemic steroid therapy (>10mg/day prednisone or equivalent) or any other form of immunosuppressive therapy, and continued to be used within 2 weeks before the first dose in this study;
* Those with multiple factors affecting oral drugs (such as inability to swallow, post gastrointestinal resection, chronic diarrhea and intestinal obstruction, etc.);
* Imaging (CT or MRI) shows that the tumor has invaded or unclearly separated the large blood vessels;
* Patients with active bleeding, or unexplained persistent decline in hemoglobin should postpone their screening/enrollment until the bleeding stops and the investigator judges it to be safe;
* Within 4 weeks before the first dose in this study, patients with CTCAE5.0 grade 3+ bleeding; patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin or their analogues; on the premise that the international normalized ratio of prothrombin time (INR) ≤1.5, it is allowed to use low-dose warfarin (≤1mg/D), low-dose heparin (≤12000U /D) or low-dose aspirin (≤100mg/D) for preventive purposes;
* Within 4 weeks before the first dose in this study, patients with unhealed wounds, fractures, gastric and duodenal active ulcers, ulcerative colitis, or unresected tumors have active bleeding, or may be caused as determined by the researchers other conditions of gastrointestinal bleeding and perforation, have undergone major surgery (excluding vascular access surgery), inoculated with preventive vaccine or attenuated vaccine;
* Received the treatment of proprietary Chinese medicines with anti-tumor indications specified in the NMPA approved drug instructions within 2 weeks before the start of the study treatment(Including compound cantharidin capsules, Kangai injection, Kanglaite capsule/injection, Aidi injection, brucea javanica oil injection/capsule, Xiaoaiping tablet/injection, Huachansu capsule, etc.); or received drugs with immunomodulatory effects (including thymosin, interferon, and interleukin, except for local use to control pleural effusion or ascites);
* History of organ or blood transplantation;
* Patients have active diverticulitis, abdominal abscess, gastrointestinal obstruction;
* Patients with any severe and/or uncontrollable disease, including:

  1) Patients with unsatisfactory blood pressure control (systolic blood pressure>140 mmHg, diastolic blood pressure>90 mmHg); 2)Within 6 months of the first administration patients with myocardial ischemia or myocardial infarction, arrhythmia that require treatment (including QTC ≥480ms), and grade ≥2 congestive heart failure; 3) active or uncontrolled serious infection (≥CTCAE5.0 Grade 2 infection), tuberculosis patients; 4) Known clinical history of liver disease, including viral hepatitis, carriers of hepatitis b virus must be excluded from active HBV infection, i.e., HBV DNA positive (>2500 copy /mL or >500IU/mL);known hepatitis c virus infection (HCV) and HCV RNA positive (>1 x 10^3 copy /mL), or other decompensated liver disease, chronic hepatitis requires antiviral treatment; 5) HIV test positive or Syphilis Testing RPR positive; 6) Diabetes is poorly controlled (fasting blood glucose (FBG) ≥10mmol/L); 7) Urine routines suggest that urine protein is ≥++, and the 24-hour urine protein quantification is more than 1.0 g;
* Those considered by the researcher to be unsuitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
PFSR-6m | up to 6 months
  Progression-Free Survival rate at 6 months.

SECONDARY OUTCOMES:
Progression-Free Survival（PFS） | up to approximately 24 months
  PFS is defined as the time from randomization until the first documented progressive disease (PD) or death from any cause response assessment, based on Response Assessment in Neuro-Oncology (RANO) prior.
Objective Response Rate（ORR） | up to approximately 24 months
  ORR is defined as percentage of subjects confirmed complete response (CR) or partial response (PR), based on Response Assessment in Neuro-Oncology (RANO) prior to progression or any further therapy.
Overall Survival（OS） | up to approximately 24 months
  From the start of treatment to the date of death or the last follow-up.
Disease Control Rate（DCR） | up to approximately 24 months
  The DCR is defined as the proportion of subjects with CR, PR, or stable disease (SD), based on Response Assessment in Neuro-Oncology (RANO) prior.
Safety | up to approximately 24 months
  Observe any adverse events that occurred in all subjects during the clinical study and within 1 month after stopping the drug, including clinical symptoms, abnormal vital signs, and abnormalities in laboratory examinations, and record their clinical features, severity, and time of occurrence, duration, treatment methods and prognostic outcome, and determine its correlation with the study drug, based on Common Terminology Criteria for Adverse Events (CTCAE) 5.0 to assess the safety.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China